CLINICAL TRIAL: NCT05048784
Title: An Open-label, Randomized, Two-way Crossover, Bioequivalence Study in Healthy Volunteers to Compare the Pharmacokinetics of Two Different Tablets of Sotorasib
Brief Title: A Study to Compare the Pharmacokinetics of Two Different Tablets of Sotorasib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20210093
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-11

CONDITIONS: Healthy Participants
Keywords: Sotorasib; AMG 510; Bioequivalence
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence ABC (Experimental): Participants will be administered sotorasib dose A orally in the following order:
  * Treatment A - as 3 tablets (test 1)
  * Treatment B - as 8 tablets (reference)
  * Treatment C - as 3 tablets (test 2)
  Interventions: Drug: Sotorasib
- Treatment Sequence BAC (Experimental): Participants will be administered sotorasib dose A orally in the following order:
  * Treatment B - as 8 tablets (reference)
  * Treatment A - as 3 tablets (test 1)
  * Treatment C - as 3 tablets (test 2)
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Oral tablet
  Other Names: AMG 510

SUMMARY:
The primary objective of this study is to compare the pharmacokinetics (PK) of sotorasib dose A administered orally as 3 tablets (test) to sotorasib dose A administered orally as 8 tablets (reference).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants or female participants, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 30 kg/m^2 (inclusive), at the time of Screening.
* Females of nonchildbearing potential.

Exclusion Criteria:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease, including history of myolysis, not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 145 participants were enrolled in the study in the United States between 16 August 2021 and 18 February 2022.
Pre-assignment Details: After randomization, participants received Treatment A (test 1) and Treatment B (reference) according to the treatment sequence assigned. A group of participants from both arm proceeded to receive Treatment C (test 2) with a high-fat meal. Dose administration of sotorasib occurred on Day 1 (Period 1) and Day 4 (Period 2) under fasted conditions and on Day 7 (Period 3) under fed condition.
Groups:
- Treatment Sequence AB: Participants were administered 960 mg sotorasib orally in the following order:
  * Period 1: Treatment A as 3 tablets (test 1).
  * Period 2: Treatment B as 8 tablets (reference).
- Treatment Sequence BA: Participants were administered 960 mg sotorasib orally in the following order:
  * Period 1: Treatment B as 8 tablets (reference).
  * Period 2: Treatment A as 3 tablets (test 1).
- Treatment Sequence ABC: Participants were administered 960 mg sotorasib orally in the following order:
  * Period 1: Treatment A as 3 tablets (test 1).
  * Period 2: Treatment B as 8 tablets (reference).
  * Period 3: Treatment C as 3 tablets with a high-fat meal (test 2).
- Treatment Sequence BAC: Participants were administered 960 mg sotorasib orally in the following order:
  * Period 1: Treatment B as 8 tablets (reference).
  * Period 2: Treatment A as 3 tablets (test 1).
  * Period 3: Treatment C as 3 tablets with a high-fat meal (test 2).
Period: Period 1
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC
Started | 66 | 66 | 6 | 7
Administered Treatment A | 66 | 0 | 6 | 0
Administered Treatment B | 0 | 66 | 0 | 7
Completed | 63 | 65 | 6 | 7
Not Completed | 3 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC
Started | 63 | 65 | 6 | 7
Administered Treatment A | 0 | 65 | 0 | 7
Administered Treatment B | 63 | 0 | 6 | 0
Completed | 63 | 64 | 6 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC
Started | 0 (Participants assigned to treatment sequence AB did not enter Period 3, as pre-specified.) | 0 (Participants assigned to treatment sequence BA did not enter Period 3, as pre-specified.) | 6 | 7
Administered Treatment C | 0 | 0 | 6 | 7
Completed | 0 | 0 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of sotorasib and had at least 1 postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence AB | Treatment Sequence BA | Treatment Sequence ABC | Treatment Sequence BAC | Total
Number analyzed (Participants) | 66 | 66 | 6 | 7 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 66 | 6 | 7 | 145
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 1 | 1 | 15
  Male | 59 | 60 | 5 | 6 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 31 | 4 | 1 | 63
  Not Hispanic or Latino | 39 | 35 | 2 | 6 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 26 | 30 | 0 | 4 | 60
  White | 39 | 34 | 6 | 3 | 82
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sotorasib for Treatments A and B
Description: Blood samples were collected by venipuncture or cannulation for measurement of plasma concentrations of sotorasib. Plasma pharmacokinetic (PK) parameters of sotorasib were summarized per treatment received, regardless of treatment sequence, as pre-specified.
Time Frame: Predose (Hour 0), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on Day 1 (Period 1) and Day 4 (Period 2)
Population: The PK population included all participants who received at least 1 dose of sotorasib in Periods 1 and 2, and had evaluable PK data. A participant may have been excluded from the PK summary statistics and statistical analysis if the participant had an adverse event (AE) of vomiting that occurred at or before 2 times median time of the Cmax (tmax) or diarrhea within 24 hours of dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: One administration of 960 mg sotorasib administered orally as 3 tablets (test 1) in Period 1 or Period 2, depending on treatment sequence assigned.
- Treatment B: One administration of 960 mg sotorasib administered orally as 8 tablets (reference) in Period 1 or Period 2, depending on treatment sequence assigned.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 142 | 141
ng/mL | 6650 (41.3) | 6540 (37.3)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Statistical analysis was conducted to investigate the bioequivalence of treatment A (test 1) to treatment B (reference) for Cmax; Ratio of geometric least squares means = 1.009, 90% CI 2-sided [0.980 to 1.040] — The geometric least squares mean ratios and confidence intervals (Cls) were obtained by taking the exponential of the corresponding differences and Cls on the natural-log (In) scale

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Sotorasib for Treatments A and B
Description: Blood samples were collected by venipuncture or cannulation for measurement of plasma concentrations of sotorasib. Plasma PK parameters of sotorasib were summarized per treatment received, regardless of treatment sequence, as pre-specified.
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least 1 dose of sotorasib in Periods 1 and 2, and had evaluable PK data. A participant may have been excluded from the PK summary statistics and statistical analysis if the participant had an AE of vomiting that occurred at or before 2 times median tmax or diarrhea within 24 hours of dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 142 | 140
h*ng/mL | 27800 (51.1) | 27500 (41.6)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Statistical analysis was conducted to investigate the bioequivalence of treatment A (test 1) to treatment B (reference) for AUClast; Ratio of geometric least squares means = 1.010, 90% CI 2-sided [0.967 to 1.055] — The geometric least squares mean ratios and Cls were obtained by taking the exponential of the corresponding differences and Cls on the In scale

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Sotorasib for Treatments A and B
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 138 | 138
h*ng/mL | 28600 (48.1) | 27700 (41.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Statistical analysis was conducted to investigate the bioequivalence of treatment A (test 1) to treatment B (reference) for AUCinf; Ratio of geometric least squares means = 1.020, 90% CI 2-sided [0.977 to 1.065] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent AE (TEAE)
Description: An AE is any untoward medical occurrence in a participant irrespective of a causal relationship with the study treatment.
  Any abnormal clinical laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., 12-lead electrocardiogram or vital signs measurements), including those that worsen from baseline, that are considered clinically significant in the medical and scientific judgment of the Investigator (i.e., not related to progression of underlying disease) were considered AEs.
Time Frame: Day 1 to Day 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Treatment C: One administration of 960 mg sotorasib administered orally as 3 tablets with a high-fat meal (test 2) in Period 3.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 145 | 145 | 13
Participants | 8 | 10 | 0

5. Secondary Outcome: Food Effect: Cmax of Sotorasib
Description: Blood samples were collected by venipuncture or cannulation for measurement of plasma concentrations of sotorasib.
Time Frame: Predose (Hour 0), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on Day 1 (Period 1), Day 4 (Period 2), and Day 7 (Period 3)
Population: The PK population included all participants who received at least 1 dose of sotorasib in Period 3 and had evaluable PK data. A participant may have been excluded from the PK summary statistics and statistical analysis if the participant had an AE of vomiting that occurred at or before 2 times median tmax or diarrhea within 24 hours of dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 13
ng/mL | 6390 (34.6) | 6790 (28.9) | 6400 (19.0)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other — Statistical analysis was conducted to investigate the food effect of treatment C (test 2) to treatment A (test 1) for Cmax; Ratio of geometric least squares means = 1.001, 90% CI 2-sided [0.836 to 1.199] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Food Effect: AUClast of Sotorasib
Description: Blood samples were collected by venipuncture or cannulation for measurement of plasma concentrations of sotorasib.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 13
h*ng/mL | 23900 (40.8) | 26100 (31.1) | 34500 (19.2)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other — Statistical analysis was conducted to investigate the food effect of treatment C (test 2) to treatment A (test 1) for AUClast; Ratio of geometric least squares means = 1.447, 90% CI 2-sided [1.200 to 1.745] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Food Effect: AUCinf of Sotorasib
Description: Blood samples were collected by venipuncture or cannulation for measurement of plasma concentrations of sotorasib.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 12 | 13 | 13
h*ng/mL | 23500 (41.0) | 26500 (30.3) | 34700 (19.2)
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Other — Statistical analysis was conducted to investigate the food effect of treatment C (test 2) to treatment A (test 1) for AUCinf; Ratio of geometric least squares means = 1.484, 90% CI 2-sided [1.236 to 1.783] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 9
Description: The safety population included all participants who received at least 1 dose of sotorasib and had at least 1 postdose safety assessment.
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/145 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/145 | 0/13
Other Adverse Events (participants affected / at risk) | 8/145 | 10/145 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=145) | Treatment B (N=145) | Treatment C (N=13)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT05048784/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT05048784/SAP_001.pdf